CLINICAL TRIAL: NCT01635530
Title: Study of Lyme Neuroborreliosis: Epidemiology, Manifestations, Diagnostics and Treatment
Brief Title: Study of Lyme Neuroborreliosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Jarmo Oksi, vs.prof, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T1/2012
Record Dates: First submitted 2012-07-03; First posted 2012-07-09 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Lyme Neuroborreliosis
Keywords: doxycycline; ceftriaxone
MeSH Terms: conditions — Lyme Neuroborreliosis | interventions — Doxycycline; Ceftriaxone

ARMS (2):
- Ceftriaxone (Active Comparator): Treatment of intravenous ceftriaxone (2 g/day), three weeks
  Interventions: Drug: Ceftriaxone
- Doxycycline (Experimental): Treatment with oral doxycycline (200mg / day), four weeks
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Doxycycline — Doxycycline: 100mg tablet two times per day, four weeks
  Arms: Doxycycline
Drug: Ceftriaxone — 2 g intravenous once a day, three weeks
  Arms: Ceftriaxone

SUMMARY:
The main purpose of this study is to determine whether four weeks treatment with oral doxycycline is as equally effective as three weeks treatment with intravenous ceftriaxone in patients with Lyme neuroborreliosis. The other purpose is to improve laboratory diagnostics of Lyme neuroborreliosis and further define the manifestations and epidemiology of the disease in Finland.

ELIGIBILITY:
Inclusion Criteria for definite Lyme neuroborreliosis (Criteria 1-3 or 1 and 4 fulfilled):

1. Neurological symptoms suggestive of LNB without other obvious reasons
2. CSF pleocytosis (>4 leukocytes per mikrol)
3. Intrathecal production of B. burgdorferi specific antibodies
4. Detection of B. burgdorferi DNA in central spinal fluid

Inclusion Cirteria for possible LNB (criteria 1 and 2 or 3 fullfilled):

1. Neurological symptoms suggestive of LNB wihtout other obvious reasons
2. Production of B. burgdorferi spesific antibodies in serum
3. Erythema migrans during the previous three months

Exclusion Criteria:

* pregnancy and breastfeeding
* women planning to get pregnant in two months
* age under 18
* handicapped persons
* prisoners
* use of any antibiotics two weeks before study treatments begins
* allergy for tetracyclines or cephalosporins

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
The improvement of the clinical condition during the study. | 12 months
  The clinical condition of participants will be evaluated with visual analogue scale (from 0 to 10, 0=best) by the participants. The VAS scores are collected before the treatment with antibiotics, and 4 months and 12 months after the treatment.
The clinical condition evaluated by the participants after 12 months from the treatment | 12 months
  The clinical condition is evaluated with VAS by the participants.

SECONDARY OUTCOMES:
Central spinal fluid (CSF) pleocytosis | 3 weeks
  The decline in CSF leukocyte count between the patients in doxycycline and ceftriaxone groups
CSF protein concentration | 3 weeks
  The decline in CSF protein concentration between the patients in doxycycline and ceftriaxone groups.
CSF lactate level | 3 weeks
  The decline in CSF lactate level between the patients in doxycycline and ceftriaxone groups.
CSF CXCL13 concentration | 3 weeks
  The decline in CSF CXCL13 concentration wetween the patients in doxycycline and ceftriaxone groups

CONTACTS AND LOCATIONS:
Overall Officials: Jukka Hytönen, Principal Investigator — University of Turku; Elisa Kortela, Principal Investigator — HYKS; Mari Kanerva, Principal Investigator — HYKS; Laura Airas, Principal Investigator — TYKS
Locations (2):
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Turku University Hospital, Turku

REFERENCES:
- [Derived] Kortela E, Kanerva MJ, Puustinen J, Hurme S, Airas L, Lauhio A, Hohenthal U, Jalava-Karvinen P, Nieminen T, Finnila T, Haggblom T, Pietikainen A, Koivisto M, Vilhonen J, Marttila-Vaara M, Hytonen J, Oksi J. Oral Doxycycline Compared to Intravenous Ceftriaxone in the Treatment of Lyme Neuroborreliosis: A Multicenter, Equivalence, Randomized, Open-label Trial. Clin Infect Dis. 2021 Apr 26;72(8):1323-1331. doi: 10.1093/cid/ciaa217. PMID 32133487